CLINICAL TRIAL: NCT00999895
Title: A Non-interventional, Prospective, Open-label Study for the Evaluation of the Selection and Outcome of the Antipsychotic Treatment Switch in Outpatients With Schizophrenia - ETOS Study
Brief Title: A Study Evaluating the Treatment Selection and Outcome When Changing Antipsychotic Treatment in Schizophrenic Patients
Acronym: ETOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NGR-DUM-2009/1
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Switch of antipsychotic treatment; Outcome evaluation; monotherapy; Greece
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Antipsychotic outpatients with schizophrenia: Switched treatment of antipsychotic outpatients with schizophrenia

SUMMARY:
The purpose of the study is to evaluate the outcome of treatment switch defined as an improvement in CGI-CB scale (Clinical Global Impression - Clinical Benefit).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (as per DSM-IV), at least 6 months prior to enrolment in the study
* Subjects who have initiated a new antipsychotic treatment within the preceding 2 weeks
* Subjects whose prior and current antipsychotic treatment consists of any typical or atypical antipsychotic monotherapy

Exclusion Criteria:

* Subjects fulfilling criteria for diagnosis of any other psychiatric condition (except from schizophrenia), as per DSM-IV Axis Ι, concomitant organic mental disorder or mental retardation
* Substance abuse or dependence (with the exception of nicotine dependence), as defined by DSM-IV criteria and not in full remission
* Female subjects who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone a switch in their antipsychotic treatment and fulfill the following criteria will participate in the study.
Sampling Method: Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
CGI-CB scale score of subjects achieving a score of < 4. | At Week 18 - once

SECONDARY OUTCOMES:
Change in PANSS scale | Baseline (Day 0) to the end of study treatment (week 6, week 12, week 18) or the premature study withdrawal of the subject - up to 4 times in 18 weeks
Change in BARS scale | Baseline (Day 0) to the end of study treatment (week 6, week 12, week 18) or the premature study withdrawal of the subject - up to 4 times in 18 weeks
Changes in CGI-S and CGI-I scales | Baseline (Day 0) to the end of study treatment (week 6, week 12, week 18) or the premature study withdrawal of the subject - up to 4 times in 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, Dr., Study Director — Marketing Company Medical and Regulatory Affairs Director, AstraZeneca S.A. Greece
Locations (43):
- Greece (43):
  - Research Site, Pátrai, Achaias
  - Research Site, Nafplion, Argolidas
  - Research Site, Tripoli, Arkadias
  - Research Site, Athens, Attica
  - Research Site, Dafni, Attica
  - Research Site, Drapetsona, Attica
  - Research Site, Exarcheia, Attica
  - Research Site, Glifada, Attica
  - Research Site, Ilioúpoli, Attica
  - Research Site, Ilissia, Attica
  - Research Site, Koridalos, Attica
  - Research Site, Marousi, Attica
  - Research Site, N. Makri, Attica
  - Research Site, P. Faliro, Attica
  - Research Site, Pangrati, Attica
  - Research Site, Peristeri, Attica
  - Research Site, Petroúpolis, Attica
  - Research Site, Piraeus, Attica
  - Research Site, Zografos, Attica
  - Research Site, Athens, Attikis
  - Research Site, Koropí, Attikis
  - Research Site, Néo Irákleio, Attikis
  - Research Site, Chania, Chanion
  - Research Site, Kos, Dodekanissou
  - Research Site, Corfu, Eptanisa
  - Research Site, Agrinio, Etoloakarnanias
  - Research Site, Alexandroupoli, Evrou
  - Research Site, Lamia, Fthiotidos
  - Research Site, Heraklio, Herakliou
  - Research Site, Véroia, Imatheias
  - Research Site, Ioannina, Ioanninon
  - Research Site, Karditsa, Karditsas
  - Research Site, Kavala, Kavalas
  - Research Site, Larissa, Larissas
  - Research Site, Volos, Magnisias
  - Research Site, Kalamata, Mesinias
  - Research Site, Giannitsá, Pellas
  - Research Site, Rethymno, Rethimnou
  - Research Site, Komotini, Rodopis
  - Research Site, Serres, Serres
  - Research Site, Thessaloniki, Thessalonikis
  - Research Site, Trikala, Trikalon
  - Research Site, Thebes, Viotias

REFERENCES:
- [Derived] Roussidis A, Kalkavoura C, Dimelis D, Theodorou A, Ioannidou I, Mellos E, Mylonaki T, Spyropoulou A, Yfantis A. Reasons and clinical outcomes of antipsychotic treatment switch in outpatients with schizophrenia in real-life clinical settings: the ETOS observational study. Ann Gen Psychiatry. 2013 Dec 20;12(1):42. doi: 10.1186/1744-859X-12-42. PMID 24359635